CLINICAL TRIAL: NCT02745275
Title: Supporting Healthy Aging by Peer Education and Support (SHAPES) - A Stepped-Wedge Cluster Randomized Trial
Brief Title: Supporting Healthy Aging by Peer Education and Support
Acronym: SHAPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Covenant Health, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: SHAPES-0915
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Health Behavior; Ageing
Keywords: Peer Education; Health Coaches; Community Dwelling Seniors; Health Literacy; Health Education; Healthy Ageing
MeSH Terms: conditions — Health Behavior; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-led Health Education (Experimental): A single 60 minute interactive workshop led by the trained health coach followed by a series of three one hour discussion groups
  Interventions: Behavioral: Peer-led Health Education
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Peer-led Health Education — Peer-led health education
  Arms: Peer-led Health Education

SUMMARY:
Canadians are living longer than ever before. However, many in our society age with long term chronic medical conditions which have a major impact on their need for healthcare, their quality of life and well-being. Encouragement of lifestyle practices which promote healthy aging and self-management techniques to deal with chronic disease is important in improving peoples' well-being

The purpose of this study is to study the impact of peer delivered education and support for seniors living in the community to see if training given to other seniors improves healthy ageing behaviours and their health literacy.

DETAILED DESCRIPTION:
In Canada, between 1960 and 2009, the proportion of seniors (people aged ≥65 years) rose from 8% to 14%; it is estimated that this proportion will increase to 23-25% by 2036. The number of people in the population aged ≥80 years is projected to more than double between 2009 and 2036. This population ageing has, and will, have a major impact on healthcare, economics, education, employment and social engagement. Many in our society age with long term chronic medical conditions; the management of which is partly responsible for the increasing consumption of health care resources in later life. There is a pressing need on the part of health care providers and policy makers to contain these increasing expenditures. Encouragement of lifestyle practices which promote successful or healthy aging and self - management techniques to deal with chronic disease are therefore of paramount importance to the achievement of this goal. Cost containment, however, is not the sole reason for pursuing such practice; there is some evidence that self-management and an increase in health literacy leads to an increased sense of empowerment and an improvement in health related quality of life for seniors.

In the presence of chronic disease, self-management is seen as a critical element in containing resource demand and in empowering patients whilst increasing their health literacy. Self-management training courses have been developed for generic physical long term conditions which have led to improved outcomes and some cost savings in chronic care. There is therefore an opportunity to educate and empower seniors in both healthy ageing behaviours and self-management of chronic disease, which has the potential to contain health care resource use, improve perception of self-rated health and quality of life.

This study aims to explore the use of health coaches, where health coaching can be defined as helping patients gain the knowledge, skills, tools and confidence to become active participants in their care so that they can reach their self-identified health goals, drawn from community dwelling seniors, rather than "expert patients" in educating and supporting their peers in healthy aging behaviours and self-management of chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female community dwelling seniors who attend seniors centres in Edmonton
* Able to commit their time to participate in the study and complete the required assessments
* Speak and understand English
* Be under the care of or have access to a Family doctor

Exclusion Criteria:

* Medical or psychological impairment which might seriously impair adherence to the program

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Self-Rated Abilities for Healthy Practices Scale | 18 months
  Change in proportion of participating seniors engaged in healthy aging behaviours following the intervention compared to unexposed controls

SECONDARY OUTCOMES:
Change in physical activity levels measured by the Physical Activity Scale for the Elderly (PASE) | 12 months
Number of participants seeking health care as measured by Health care seeking and resource use questionnaire | 12 months
Measure self-efficacy for participating seniors using The General Self-Efficacy Scale (GES) | 12 months
Participant's willingness to change assessed by readiness to change ruler | 12 months
Number of participating seniors satisfied with the health coaches assessed by a semi-structured interviews | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian S Wagg, MD, Principal Investigator — University of Alberta
Locations (1):
- Division of Geriatric Medicine, Clinical Sciences Building, University of Alberta Hosp, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Foster G, Taylor SJ, Eldridge SE, Ramsay J, Griffiths CJ. Self-management education programmes by lay leaders for people with chronic conditions. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD005108. doi: 10.1002/14651858.CD005108.pub2. PMID 17943839
- [Background] Bodenheimer T, Lorig K, Holman H, Grumbach K. Patient self-management of chronic disease in primary care. JAMA. 2002 Nov 20;288(19):2469-75. doi: 10.1001/jama.288.19.2469. PMID 12435261
- [Background] Fiocco AJ, Scarcello S, Marzolini S, Chan A, Oh P, Proulx G, Greenwood C. The effects of an exercise and lifestyle intervention program on cardiovascular, metabolic factors and cognitive performance in middle-aged adults with type II diabetes: a pilot study. Can J Diabetes. 2013 Aug;37(4):214-219. doi: 10.1016/j.jcjd.2013.03.369. Epub 2013 Aug 2. PMID 24070883
- [Background] Lorig KR, Sobel DS, Stewart AL, Brown BW Jr, Bandura A, Ritter P, Gonzalez VM, Laurent DD, Holman HR. Evidence suggesting that a chronic disease self-management program can improve health status while reducing hospitalization: a randomized trial. Med Care. 1999 Jan;37(1):5-14. doi: 10.1097/00005650-199901000-00003. PMID 10413387